

# Clinical Investigation Plan

U009

Safety and performance of short- and long-term Baseplates

for attaching the Marco Recorder

(Brand name: UNEEG Episight)

September 2021 - December 2022

2022-06-16 Page 1 of 4



#### SYNOPSIS OF THE CLINICAL INVESTIGATION

| Safety and performance of short- and long-term Baseplates for attaching the Marco Recorder The study is divided into two parts. In the initial part (Main part/Part I) of the study, the inclusion period is up to 42 days for each subject, where the test period is divided into 2 periods of 17-18 days each. After the initial part of the study, an interim analysis will be performed and the result will be used to conduct a subsequent study period (Extension part/Part II) of up to 42 days including additional subjects. | Title | Duration |
|---|---|---|
| | term Baseplates for attaching the Marco | (Main part/Part I) of the study, the inclusion period is up to 42 days for each subject, where the test period is divided into 2 periods of 17-18 days each. After the initial part of the study, an interim analysis will be performed and the result will be used to conduct a subsequent study period (Extension part/Part II) of up to 42 days including additional |

#### Introduction

UNEEG™ medical is developing a new version of the 24/7 EEG™ SubQ system, which is used for ultra long-term ambulatory EEG recording. The current system consists of an implantable electrode and an external Recorder connected to a "disc" with a cable. The Recorder acts as a power source and data storage unit. When the disc is placed on the skin over the implant it receives a magnetic inductive link that 1) powers the electrode, and 2) transfers the recorded EEG signals to the Recorder. UNEEG™ medical is developing a new external power and storage unit with the in-house development name "Marco Recorder", which is a smaller and cable-free replacement of the current version. The new Recorder is attached to the skin behind the ear by mounting it in a Baseplate consisting of a double adhesive and a plastic frame.

The purpose of this clinical investigation is to test the safety and performance of short- and long-term Baseplates constructed with different types of biocompatible adhesives. The short-term Baseplate must be replaced daily and the long-term every four days. The outcome of the investigation will be used by UNEEG™ medical to evaluate two Baseplates, one short-term and one long-term Baseplate, suitable for attaching the Marco Recorder to the skin behind the ear.

# **Objective**

**The primary objective** of the study is to demonstrate the skin-friendliness of two types of Baseplates (i.e., adhesives) after up to 35 days repeated use on the skin behind the ear.

## The secondary objectives are to

- Demonstrate effectiveness of the Baseplate to hold the Recorder in place on the skin behind the ear.
- Evaluate safety of the Baseplate (i.e., adhesives).
- Evaluate subject-reported performance of the different types of Baseplates and the Recorder.
- Evaluate subject-reported satisfaction.

It is hypothesised that the various Baseplates can 1) hold a Recorder in place for 1 or up to 4 days depending on the type of adhesive, 2) be worn and removed gently without significantly irritating or damaging the skin.

## **Endpoints**

## **Primary endpoint**

The trans epidermal water loss (TEWL) is captured to evaluate skin barrier functionality, i.e. to measure potential skin damage caused by repeated use of the Baseplate and Recorder.

## Secondary endpoints



## Skin assessment endpoints

- Hydration: An objective skin assessment based on conductance to measure the skin's ability to retain water.
- Erythema: An objective skin assessment based on reflectance spectrophotometry to measure reddening.
- Pain upon removal is assessed by a Visual Analog Score (VAS) on a scale between 1-10).
- Skin condition is based on visual inspection by investigator (including a photo) and by subject -report.

# Safety endpoint

 Nature and frequency of adverse events during the study and their severity, outcomes, and relationship to the Baseplate and Recorder.

## Performance & effectiveness endpoints (subject-reported)

- Daily: Subject questionnaire on physical activity and complications with devices.
- End of each test period: Subject questionnaire on user experience.

# **User Satisfaction Endpoint**

• End of study: Subject satisfaction questionnaire.

# **Design and Methods**

The first study part (Main part/Part I) is a randomised, controlled setup with an initial 2x2 cross-over design consisting of two test periods of 17-18 days each. Thirty subjects will be included in this part, and each individual subject will test two short-term Baseplates (type A behind one ear and type B behind the other ear) in one test period (17-18 days) and two long-term Baseplates (type C and D) in a second test period of the same duration. The order of the two test periods (short/long-term Baseplate) and the site of attachment (left/right ear) will be randomised. Following this study part (Part I), an interim analysis will be performed to select the most promising short-term and long-term Baseplate (i.e., adhesive) to be tested in the Extension part/Part II with a modified design. Thus, in the second study part (Extension part/Part II) 10 additional subjects will be included to test the selected Baseplates in a randomized controlled setup for a period of 35 days.

The study will take place in Denmark at Bispebjerg Hospital.

## Population/subjects

The investigational population consists of 40 healthy subjects who comply with the following selection criteria:

#### Inclusion Criteria:

- Informed consent obtained, and letter of authority signed before any study related activities
- Are at least 18 years of age and have full legal capacity
- Have healthy skin behind the ear

#### **Exclusion Criteria:**

- Pregnant or breastfeeding<sup>1</sup>
- Known allergic responses to the adhesives
- Treatment with corticosteroids, either as a cream in the area behind the ear or systemically (tablet or injection) within the last month
- Subject is unable or does not have the necessary assistance to properly operate the device system

<sup>&</sup>lt;sup>1</sup> Pregnancy is screened for through a pregnancy test before inclusion of fertile women.



# Investigational device and comparator

The investigational devices are non-CE marked biocompatible Baseplates and a non-functional Recorder. Four different Baseplates are identified as Baseplate A, B, C and D. Type A and B are tested for short-term (daily) use, and type C and D are tested for long-term (4 days) use. All types of Baseplates are biocompatible and intended for attaching other medical devices (1–4).

# Investigation approval

The investigation will be approved by the local ethics committee (EC) and the regulatory authorities (LMS) in Denmark before initiating the investigation.